CLINICAL TRIAL: NCT03976804
Title: Epidemiological Study to Assess the Prevalence of Lung Cancer in Patients With Smocking-associated Atherosclerotic Cardiovascular Diseases
Brief Title: Epidemiological Study to Assess the Prevalence of Lung Cancer
Acronym: PREVALUNG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Centre Chirurgical Marie Lannelongue (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2019-A00262-55
Record Dates: First submitted 2019-06-03; First posted 2019-06-06 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Lung Cancer; Tobacco; Atherosclerotic Cardiovascular Event
Keywords: Cancer; Tobacco
MeSH Terms: conditions — Lung Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- atherosclerotic cardiovascular event associated with tobacco (Experimental)
  Interventions: Other: low dose CT scan; Other: blood sample collection; Other: faecal sample collection

INTERVENTIONS:
Other: low dose CT scan — Lung cancer screening will be based on the analysis of a low dose CT scan
Other: blood sample collection — establish a phenotyping of immunity, blood inflammation and digestive and tumour microbiota
Other: faecal sample collection — establish a phenotyping of immunity, blood inflammation and digestive and tumour microbiota

SUMMARY:
Lung cancer is the main cause of mortality by cancer in France. The lung cancer stage at time of diagnosis is a major determinant of survival. To date, 75% of lung cancer are diagnosed at an advanced stage with worse survival). Lung cancer screening is based on low dose CT scan which allows to decrease lung cancer related mortality of 20% in patients aged 55-74 years-old with a history of tobacco consumption ≥ 30 PY active of who quite < 15 years. These criteria for eligibility for lung cancer screening lead to 1 to 2% of lung cancer diagnosis at the first CT scan. In our experience regarding 1 year of lung cancer surgical resection, only 45% of the patients presented criteria for lung cancer screening. Moreover, the duration of tobacco consumption would provide a better stratification of lung cancer risk compared to only PY. Therefore, other criteria for lung cancer screening eligibility could be proposed. Currently, 9 out of 10 lung cancer is linked with tobacco consumption which is also a major risk factor for atherosclerosis-associated cardiovascular events. Around 40% of patients with a lung cancer have a history of atherosclerosis-associated cardiovascular event, mainly coronary artery diseases and peripheral artery diseases. Main Objective: The objective is to compare the observed rate of lung cancer prevalence in our study to the rate of around 2 % observed in lung cancer screening trials in south Europe (France and Italy).

The investigators hypothesize that the population of patients with a history of atherosclerotic cardiovascular event associated with tobacco consumption present a higher prevalence of lung cancer compared with the population of patients eligible for lung cancer screening program which is defined by age and history of tobacco consumption.

ELIGIBILITY:
Inclusion Criteria:

* Age 45 - 75 years old
* Patient who has signed an informed written consent
* Daily smoking for at least 10 years
* History of cardiovascular disease:

Exclusion Criteria:

* History of active cancer < 5 years (except in situ cervical carcinoma and basal cell carcinoma of the skin)
* Lung cancer symptoms (involuntary weight loss > 6.8 kg in 1 year, hemoptysis)
* Treatment or bleeding risk syndrome contraindicating an invasive diagnostic procedure within 3 months.
* Active pulmonary parenchymal infection
* Severe cardiac or respiratory insufficiency (resting dyspnea)

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2019-11-04 (Actual); Primary Completion 2021-05-04 (Actual); Study Completion 2022-12-02 (Estimated)

PRIMARY OUTCOMES:
prevalence of lung cancer | 19 months
  estimation of the prevalence of lung cancer among patients managed for atherosclerosis-related cardiovascular events associated with tobacco consumption.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Chirurgical Marie Lannelongue, Le Plessis-Robinson, France

REFERENCES:
- [Derived] Boulate D, Fidelle M, Caramella C, Issard J, Planche O, Pradere P, Garelik D, Hache O, Lamrani L, Zins M, Beaussier H, Chatellier G, Fadel E, Zitvogel L, Besse B, Mercier O. Epidemiological Study to Assess the Prevalence of Lung Cancer in patients with smoking-associated atherosclerotic cardiovascular diseases: PREVALUNG study protocol. BMJ Open. 2022 Dec 26;12(12):e067191. doi: 10.1136/bmjopen-2022-067191. PMID 36572501